CLINICAL TRIAL: NCT06263439
Title: Prospective Clinico-virological Surveillance of Diseases Foot-hand-mouth/Herpangina Associated With Enteroviruses in Pediatric Outpatients
Brief Title: Surveillance of HFMD in Pediatric Outpatients
Acronym: PMB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2023 MIRAND; 2023-A00585-40 (Other: ANSM)
Record Dates: First submitted 2023-06-09; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Hand, Foot and Mouth Disease; Herpangina; Enterovirus Infections
Keywords: Hand, foot and mouth disease; Enterovirus A71; Coxsackievirus A6; Herpangina; Primary care in paediatrics
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Herpangina; Enterovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Throat swab Buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with hand, foot and mouth disease or herpangina: Children with hand, foot and mouth disease or herpangina will be proposed to have a throat or buccal swab collected to do the diagnosis of an enterovirus infection.
  Interventions: Diagnostic Test: Throat/buccal swab sample

INTERVENTIONS:
Diagnostic Test: Throat/buccal swab sample — The study involves the genome detection of enteroviruses in throat or mouth swabs taken from children with a diagnosis of HFMD or herpangina. If positive, the precise type of enterovirus responsible will be identified by sequencing a viral genomic region.
  Other Names: Enterovirus genome detection (Enterovirus R-gene, bioMérieux)

SUMMARY:
The aims of this prospective multicentric study is to determine the types of enteroviruses (EVs) responsible for hand, foot and mouth disease (HFMD) or herpangina in children seen within an ambulatory setting :

* to detect an EV-A71 epidemic or another type associated with atypical forms of the disease at an early stage
* to describe and compare the epidemiological, demographic, clinical and virological characteristics of these infections between the different types of EV.

DETAILED DESCRIPTION:
Any child presenting signs suggestive of HFMD/Herpangina can be included in the study by one of the investigating paediatricians. After giving the information note to the parents (and to children over 3 years of age) and asking them not to object, the paediatrician collects a throat or mouth swab to confirm the enterovirus infection. At the same time as the swab is taken, anonymised demographic and clinical data are collected by the doctor during the consultation. The sample and the information sheet are sent to the National Reference Laboratory for enteroviruses (Clermont-Ferrand University Hospital).The diagnosis is performed by EV genome detection and if positive, genotyping is done to identify the type of the enteroviruses.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 10 years presenting with HFMD or herpangina

Exclusion Criteria:

* Refusal to participate by holders of parental authority
* Refusal to participate for children over 3 years of age

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 0 and 10 years seen for HFMD/Herpangina by one of the paediatric investigators.
  HFMD is defined by the presence of at least two of the following clinical signs:
  * a vesicular or non-vesicular rash on :
    * the palms of the hands
    * soles of the feet, or the buttocks
    * knees or elbows,
    * mouth or perioral ulcers,
  * vesicular or non-generalized eruption.
  Herpangina is defined by the presence of oral ulcers located mainly in the posterior part of the oral cavity: palate, uvula.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2028-06-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of different types of Enteroviruses | 5 years
  Prevalence of different types of enteroviruses associated with HFMD/Herpangina, determined by genomic detection of an enterovirus in samples sent to the National Reference Laboratory for enteroviruses. This will be carried out on a throat or mouth swab taken from a child seen in consultation for HFMD or herpangina at the time of the patient's inclusion in the study. Genomic detection will be carried out using real-time Reverse Transcription-Polymerase Chain Reaction, the reference method for diagnosing enterovirus infections. The type of enterovirus will then be identified by genotyping the sequence encoding the structural proteins or sequencing the complete enterovirus genome.

SECONDARY OUTCOMES:
Clinical characteristics of HFMD/Herpangina according to the different types of enteroviruses | 5 years
  Comparison between types of enteroviruses determined by genomic detection and clinical characteristics of HFMD/Herpangina. These are collected by the pediatrician during the consultation and include: the nature (throat or mouth) and the date of the sample, the date of onset of the illness, fever, the type and location of rashes, oral ulcerations or perioral, herpangina as well as digestive, ENT, respiratory, neuro-meningeal or other signs (specifying).

CONTACTS AND LOCATIONS:
Overall Officials: Audrey MIRAND, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No